CLINICAL TRIAL: NCT06736132
Title: Comparison of Different Oxygen Flow Rates During Preoxygenation Using High-Flow Nasal Oxygen
Acronym: PREFLOW2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Albin Sjöblom, Principal Investigator, Region Stockholm
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNR: 2024-04565-01; SLS-1000363 & SLS-999871 (Other Grant/Funding Number: Läkaresällskapet)
Record Dates: First submitted 2024-12-09; First posted 2024-12-16 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2024-12

CONDITIONS: Airway Anesthesia; Preoxygenation; High Flow Nasal Canula
Keywords: Preoxygenation; High-flow nasal oxygen; Anaesthesia induction

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High-flow nasal oxygen, flow rate 45 l/min (Active Comparator): Preoxygenation using high-flow nasal oxygen with a flow rate of 45 l/min
  Interventions: Device: High-flow nasal oxygen
- High-flow nasal oxygen, flow rate 70 l/min (Experimental): Preoxygenation using high-flow nasal oxygen with a flow rate of 70 l/min
  Interventions: Device: High-flow nasal oxygen
- High-flow nasal oxygen, flow rate 95 l/min (Experimental): Preoxygenation using high-flow nasal oxygen with a flow rate of 95 l/min
  Interventions: Device: High-flow nasal oxygen

INTERVENTIONS:
Device: High-flow nasal oxygen — In this study, we will use high-flow nasal oxygen for preoxygenation in patients undergoing elective anaesthesia. Preoxygenation with high-flow nasal oxygen is most often performed at flow rates of <50 l/min. In this study, patients will be randomised to preoxygenation using high-flow nasal oxygen and flow rates of 45 l/min, 70 l/min or 95 /min.

SUMMARY:
High-flow nasal oxygen (HFNO) has been used for many years to help people with breathing difficulties in the intensive care and after surgery. More recently, it has become a helpful tool during induction of anaesthesia to prevent oxygen levels from dropping when managing the airway. HFNO is particularly effective at delivering oxygen even when a patient is not breathing (apnoea), making it useful during surgeries on the voice box (larynx) because it eliminates the need for a breathing tube, giving surgeons a clear view.

HFNO is now also being used to prepare patients for anaesthesia (preoxygenation). Research shows that it works just as well as traditional tight-fitting oxygen masks while offering added benefits like better comfort for patients, easier handling for anaesthetists, and a smooth transition to oxygen delivery during apnoea.

One reason HFNO is effective is that it creates a mild pressure in the lungs, called positive end-expiratory pressure (PEEP), which improves oxygen storage in the lungs. This pressure depends on the flow rate of oxygen and is higher when the patient keeps their mouth closed. For every increase of 10 liters per minute in flow rate, HFNO generates 1 cmH2O of PEEP. This pressure helps increase the lung's capacity to hold oxygen, making the process of preoxygenation more efficient.

Most studies on HFNO for preoxygenation have used flow rates of up to 60 liters per minute. However, we don't yet know if higher flow rates could further improve preoxygenation or extend the time patients can safely go without breathing.

DETAILED DESCRIPTION:
High-flow nasal oxygen (HFNO) has long been employed to address respiratory distress in both the intensive care unit and post-anaesthesia unit. Over the past decade, HFNO has emerged as a valuable tool for preventing oxygen desaturation during airway management in the operating theatre. Notably, HFNO demonstrates effectiveness in oxygenating patients during extended periods of apnoea, providing a reliable method for apnoeic oxygenation. This technique serves as an alternative to mechanical ventilation in laryngeal surgical procedures, offering potential advantages such as a clear operating field for surgeons without the interference of a tracheal tube.

More recently, HFNO has found application in preoxygenation before anaesthesia induction. Studies indicate that the preoxygenation efficacy of HFNO is comparable to that of a standard tight-fitting facemask, with added benefits including enhanced patient comfort, improved ease of use as assessed by anaesthetists, and the potential for a seamless transition to apnoeic oxygenation.

One of the suggested mechanisms contributing to the favourable outcomes observed with HFNO in managing patients with respiratory distress is a flow-dependent positive end-expiratory pressure (PEEP) effect. When patients breathe with a closed mouth, HFNO appears to generate a PEEP effect of 1 cmH2O for every 10 l.min-1 of flow. Prior data has demonstrated that an elevated PEEP leads to a greater functional residual capacity (FRC) and improved preoxygenation effectiveness.

Previous studies investigating HFNO for preoxygenation have used flow rates ≤ 60 l.min-1. Consequently, the impact of higher flow rates on preoxygenation effectiveness and the extension of safe apnoea time remains uncertain.

In this randomised prospective study, we aim to investigate the effectiveness of preoxygenation from HFNO using different flow rates. Seventy-five patients (25 per group) scheduled for elective surgery at the Karolinska University Hospital, will be recruited. After a signed consent, the subject will be enrolled and randomised to preoxygenation using HFNO at flow rates of 45 l/min, 70 l/min or 95 l/min.

Routine perioperative monitoring, such as peripheral oxygen saturation (SpO2) and non-invasive blood pressure will be performed. Preoperatively, an arterial catheter will be inserted. An arterial blood gas will be attained before preoxygenation for base line data regarding PaCO2, PaO2 and pH.

To enable lung impedance measurement, all subjects will be applied an appropriately sized circumferential 16-electrode belt around the torso between the fourth and sixth intercostal spaces.

Patients will be positioned supine with the head elevated at 15 degrees. All groups will undergo preoxygenation using HFNO with the flow rate determined by the randomisation. All groups will be preoxygenated for 3 minutes using 100% oxygen and closed-mouth breathing. Immediately prior to anaesthesia induction, patients will evaluate the level of discomfort of preoxygenation. Thereafter, anaesthesia is induced.

Preoxygenation will be administered to all patients until the onset of apnoea, at which point oxygen delivery via HFNO will be immediately discontinued. The patient will then undergo intubation, with apnoea maintained until their oxygen saturation drops to 93%. Once this threshold is reached, mechanical ventilation with 100% oxygen will be initiated.

ELIGIBILITY:
Inclusion Criteria:

* Adult, 18-84 years old
* ASA 1-3
* BMI < 35
* Planned for elective surgery

Exclusion Criteria:

* Cardiac disease (ischemic heart disease, heart failure (NYHA ≥2), ongoing arrhythmias, pulmonary hypertension)
* Severe asthma, moderate to severe COPD
* Pregnancy
* Smokers or former smoker last finished 1 year before inclusion
* Baseline oxygen saturation < 95%
* Nasal obstruction
* Known or anticipated difficult airway
* Patients with electrical active implants where lung impedance analysis is contraindicated
* Not capable of understanding study information and signing a written consent

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safe apnoea time | From start of apnoea after anaesthesia induction until peripheral oxygen saturation drops to 93%. This time fram will probably be between 5 and 15 minutes.
  Comparison of the time from start of apnoea until reaching a SpO2 = 93% between the different flow rates

SECONDARY OUTCOMES:
Tolerance of 360 seconds of apnoea | From apnoea start until 5 minutes of apnoea
  Comparison between the three groups of the proportion of patients tolerating 360 seconds of apnoea
Arterial oxygen levels during preoxygenation | From start of preoxygenation until end of preoxygenation (approximately 3 to 4 minutes)
  Comparison between the groups in PaO2 at 1 minute and 2 minutes of preoxygenation and at the start of apnoea
Discomfort assessment | From start of preoxygenation until the end of preoxygenation, this time fram will be three minutes.
  Comparision between the groups in the level of discomfort during preoxygenation. Discomfort will be assessed on a scale from 1 to 10 (0 = no discomfort, 10 = maximal discomfort)
Lung impedance changes | From start of preoxygenation until end of apnoea (approximately 5 to 15 minutes)
  Lung impedance measurement will be conducted before preoxygenation (baseline) after three minutes of pre-oxygenation and at the end of apnoea. Comparisons of these values, at the different time points, will be conducted between the three groups.

OTHER OUTCOMES:
Differences in end-tidal and arterial carbon dioxide levels | From start of apnoea until end of apnoea (approximately 5 to 10 minutes)
  Exploratory outcome. Describe the differences in end-tidal and arterial carbon dioxide levels immediately following termination of apnoea.
Rate of arterial carbon dioxide increase during apnoea | From start of apnoea until end of apnoea (approximately 5 to 10 minutes)
  Exploratory outcome. We will investigate the rate of increase in arterial carbon dioxide levels during the apnoeic period.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on request from the corresponding author. The data are not publicly available because they contain information that could compromise the privacy of research participants.

REFERENCES:
- [Derived] Sjoblom A, Hoffman F, Hedberg M, Forsberg IM, Jonsson Fagerlund M. Preoxygenation with high-flow nasal oxygen at various flow rates in elective surgical patients: a prospective, randomised, single-blind clinical trial. Br J Anaesth. 2025 Dec 18:S0007-0912(25)00816-5. doi: 10.1016/j.bja.2025.11.017. Online ahead of print. PMID 41419379